CLINICAL TRIAL: NCT01258218
Title: Accent MRI Pacemaker and Tendril MRI Lead New Technology Assessment
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-10-027-EU-LV
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Accent MRI Group
  Interventions: Device: Implantation of an Accent MRI device

INTERVENTIONS:
Device: Implantation of an Accent MRI device — Implantation of an Accent MRI device

SUMMARY:
The intent of this study is to evaluate the performance of the implanted Accent MRI TM system in a clinical setting and optionally in the MRI environment. This system includes the St. Jude Medical Tendril MRI™ lead and SJM Accent MRITM DR pacemaker. Also the MRI Activator™ will be evaluated in this study. The MRI Activator is a handheld device that allows the user to enable and disable MRI Settings as well as check the status of MRI Settings in the pacemaker. The patient population under study includes patients with a standard bradycardia pacing indication.

ELIGIBILITY:
Inclusion Criteria:

* Approved Class I or Class II indication per ESC guidelines for implantation of a dual chamber pacemaker or single chamber pacemaker.
* Receiving a new Accent MRITM pacemaker and Tendril MRI™ lead (either initial implant or complete system change out with no abandoned devices).
* Ability to provide informed consent for study participation.
* Is willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

Exclusion Criteria:

* Have an existing pacemaker or ICD (abandoned devices and/or leads are not allowed. A new pacemaker and lead or complete system change out is required for enrollment).
* Have an existing active/inactive implanted medical device (e. g., Neurostimulator, infusion pump, etc.).
* Have a non-MRI compatible device or material implant (e.g., intracranial aneurysm clip, non-MRI compatible devices or material, metals or alloys, etc.).
* Have a lead extender or adaptor.
* Have a mechanical, prosthetic or bioprosthetic tricuspid heart valve.
* Have an abdominal diameter (approximately > 60cm) which results in contact with the magnet façade.
* Are currently participating in a study that includes an active treatment arm.
* Are pregnant or planning to become pregnant during the duration of the study.
* Have a life expectancy of less than 6 months due to any condition.
* Are less than 18 years of age.
* Are unable to comply with the follow up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with approved Class I or Class II indication per ESC guidelines for implantation of a dual chamber pacemaker or single chamber pacemaker.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Graz, Austria